CLINICAL TRIAL: NCT00772707
Title: A 30 Day, Multi-Centered, Open Label Study To Determine Comfort and Overall Contact Lens Wearing Experience Using OPTI-FREE RepleniSH® MPDS as Compared to COMPLETE®MPS Easy Rub™ or ReNu MultiPlus® in Daily Wear Soft Contact Lens Patients
Brief Title: A Multi-Center Investigation of Patient Acceptability of OPTI-FREE RepleniSH® Multi-Purpose Disinfecting Solution (MPDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-08-14
Record Dates: First submitted 2008-10-07; First posted 2008-10-15 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-08

CONDITIONS: Myopia
Keywords: contact lens solution; OPTI-FREE RepleniSH; contact lenses
MeSH Terms: conditions — Myopia | interventions — Contact Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Opti-Free Replenish (Experimental): Multi-purpose contact lens solution for cleaning and disinfecting study contact lenses used on a daily basis for 30 days.
  Interventions: Device: Multi-Purpose Disinfecting Solution (OPTI-FREE RepleniSH); Device: Contact Lenses

INTERVENTIONS:
Device: Multi-Purpose Disinfecting Solution (OPTI-FREE RepleniSH) — OPTI-FREE RepleniSH® used according to product labeled instructions for cleaning and disinfecting study contact lenses, 30 days.
  Other Names: OPTI-FREE RepleniSH®
Device: Contact Lenses — Contact lenses per participant's habitual prescription removed nightly for cleaning and disinfecting.

SUMMARY:
The purpose of this study was to demonstrate that current successful fulltime daily wear soft contact lens wearers using competitive multi-purpose solutions will note improved comfort when using OPTI-FREE RepleniSH®.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be between 18 and 65 years of age.
2. Must wear daily wear soft contact lenses a minimum of 8 hours per day,7 days a week.
3. Must be wearing a planned replacement soft lens in a 2 week or monthly replacement modality.
4. Must be using either COMPLETE Multi-Purpose Solution (MPS) Easy Rub or ReNu MultiPlus brand solution for at least 30 continuous days prior to enrollment.
5. Must be free of any contact lens-related symptoms with regard to comfort and vision throughout their wearing hours prior to enrollment, with the exception of end-of-day dryness not limiting all day wear.
6. Must have best corrected distance visual acuity, with contact lenses, of 20/30 or better in each eye.
7. Must be willing to maintain pre-enrollment systemic medication regimens during the study.
8. Must be willing to not use any topical medications or rewetting drops during the 30 day clinical trial duration.
9. Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

1. Has used any topical medication or rewetting drops for 7 days prior to enrollment.
2. Achieves best visual correction by monovision.
3. Has modified their systemic medications within 30 days prior to enrollment.
4. Has switched brands of cosmetics during the 30 days prior to the study.
5. Has a history of allergy to any study product ingredients.
6. Is unwilling or unable to meet the study visit timeline.
7. Has any active corneal, eyelid or other anterior segment inflammation or infection, which, in the opinion of the Investigator, would adversely affect successful contact lens wear.
8. Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 US study sites.
Period: Overall Study
Arm/Group | Opti-Free Replenish
Started | 114
Completed | 111
Not Completed | 3
Not completed — Withdrawn | 3

BASELINE CHARACTERISTICS:
Arm/Group | Opti-Free Replenish
Number analyzed (Participants) | 114
Age Continuous [Mean (Full Range); unit: years] | 36 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 114

OUTCOME MEASURES:

1. Primary Outcome: Comfort Ratings at Baseline
Description: Prior to any ocular assessments at the visit, comfort ratings were collected on a questionnaire using 5-point Likert scale, with 1=Strongly Agree, 1=Agree, 3=Neutral, 4=Disagree, 5=Strongly Disagree. The percentage of participants responding with "Strongly Agree" or "Agree" for each question is presented.
Time Frame: Baseline (Day 0)
Population: 6 participants were excluded from analysis due to discontinuation of contact lens wear (1), treatment during study that might interfere with study outcome (1), withdrawal (3), and missing responses (1).
Measure: Number; unit: Percentage of Participants
Arm/Group | Opti-Free Replenish
Number analyzed (Participants) | 108
Percentage of Participants
  My lens is comfortable upon instillation | 86
  My lenses feel comfortable at the end of the day | 59
  My vision is clear at the end of the day | 57
  I am satisfied with my overall lens experience | 81

2. Primary Outcome: Comfort Ratings at 30 Days
Description: as for outcome 1
Time Frame: 30 days
Population: 5 participants were excluded from analysis due to discontinuation of contact lens wear (1), treatment during study that might interfere with study outcome (1), and withdrawal (3).
Measure: Number; unit: Percentage of Participants
Arm/Group | Opti-Free Replenish
Number analyzed (Participants) | 109
Percentage of Participants
  My lens is comfortable upon instillation | 92
  My lenses feel comfortable at the end of the day | 88
  My vision is clear at the end of the day | 91
  I am satisfied with my overall lens experience | 91
  Study product enhances wearing experience more | 71
  I will continue to use the study solution after | 81

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 1 month, 12 days.
Description: The safety population included all enrolled and exposed participants.
Arm/Group | Opti-Free Replenish
Serious Adverse Events (participants affected / at risk) | 0/114
Other Adverse Events (participants affected / at risk) | 0/114

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Alcon reserves the right of prior review of any publication or presentation of information related to the study.